CLINICAL TRIAL: NCT02479815
Title: Assessing the Safety of Iron Supplementation in Micronutrient Powder (MNPs)
Brief Title: Impact of Low Dose Iron-containing Micronutrient Powders on Iron Status and Morbidity of Young Children in Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethiopian Public Health Institute (Other Government)
Collaborators: Micronutrient Initiative (Other); Wageningen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EPHI_FSNRD_CF_MNP001
Record Dates: First submitted 2015-06-16; First posted 2015-06-24 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2017-02

CONDITIONS: Nutritional Anemia; Infant Morbidity
Keywords: Complementary feeding recommendation; Program evaluation; Process and impact evaluation; Micronutrient powder (MNP) safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1gm MNP, 15 sachets per month (Other): Quasi experimental matched control cluster design where for every child 1gm Micronutrient Powder (MNP) for two days, is given which totlas to 15 sachets per month
  Interventions: Dietary Supplement: Micronutrient Powder (MNP)

INTERVENTIONS:
Dietary Supplement: Micronutrient Powder (MNP) — Every month, 15 MNPs sachets will be provided to all children 6-23 months of age with the instruction to add them to their complementary food, to enable point-of-use fortification on every alternate day. The MNPs sachets will contain 6 mg Fe together with 14 other vitamins and minerals.

SUMMARY:
The purpose of the study is to assess the safety of iron supplementation in MNPs. A quasi-experimental matched-control cluster design will be used in, purposely selected, 18 intervention and 18 matched-control clusters of Oromia and South Nations Nationalities and People (SNNP) regions of Ethiopia. A total of 2340 infants 6-11 months of age, from intervention and non-intervention clusters will be enrolled and followed longitudinally for 12 months. Morbidity data using standardized questionnaire, will be collected at baseline, and every two weeks for a period of 12 months

Research questions to be answered in this study are:

1. Is the provision of low dose iron-containing Micronutrient Powders (MNPs) to young children with or without iron deficiency safe, as assessed by their morbidity from infectious diseases?
2. What is the impact of the provision of low dose iron-containing Micronutrient Powders (MNPs) to young children on (body) iron status? Morbidity data will be collected at baseline, and every two weeks in the same cohort of children.

Body iron status will be assessed at baseline and endline as measured by serum ferritin, serum transferrin receptor, hemoglobin concentration, CRP and AGP.

In addition data on the following outcomes will be collected in these children:

1. Anthropometry (weight, height, MUAC) every 4 months
2. Breastfeeding status and consumption of processed complementary food portions in the previous week -every 4 months
3. Compliance to study intervention.

DETAILED DESCRIPTION:
For morbidity assessment 65 eligible children per cluster (18 intervention and 18non-intervention villages) a total of 2340 will be randomly selected The sample size was calculated based on an expected 12% increase in the incidence of overall diarrhoea and 30% decrease in anemia in the intervention group. The investigators assume that the investigators will be able to detect this increase with 80% power and 95% confidence interval, with an assumed 10% drop-out and design effect of two.

* Morbidity from infectious diseases will be assessed by means of a standardized recall questionnaire. Data will be collected on the following symptoms: diarrhea, respiratory signs, fever and other illnesses. Children who require medical treatment will be examined by a Health Officer at the health center following standard protocols of the Federal Ministry of Health.
* Biochemical iron status will be assessed from non-fasting venous morning blood samples. Blood samples will be kept cool and serum separated and frozen at -20oC within 3 hours of collection. Hemoglobin, serum ferritin, C-reactive protein (CRP), soluble transferrin receptor and AGP will be assessed following standardized methodologies at the laboratories of the Ethiopian Public Health Institute (EPHI).
* Anthropometry: Trained field staff will collect duplicate measurements every four months of weight, recumbent length (infants) and height (children > 12 months) using standardized methods and high quality equipment. Z-scores for length-for-age (LAZ), weight-for-age (WAZ) and weight-for-length (WLZ) will be calculated, using the 2006 WHO Child Growth Standard; and stunting, under-weight and wasting will be defined as LAZ, WAZ and LAZ <-2 SD, respectively.
* Infant feeding status. Information on infant feeding status will be collected every four months by means of a standardized questionnaire.
* Compliance to the program intervention: will be assessed by counting the number of returned and used MNP sachets every 2 weeks.
* Social, economic and demographic characteristics: will be collected in baseline questionnaires using Demographic and Health Survey methods.

Data will be analysed on an intention-to-treat basis, using the SPSS 19.0 statistical program. Random effect models will be used to account for repeated measures or episodes within children, and multiple children in each cluster.

For morbidity, the number of actual surveillance days will be counted by subtracting the days on which no recall data were available from the total days of follow-up. For the analysis of disease incidence, differences between groups will be assessed with random effects regression including number of episodes as dependent, control- or intervention as independent, and total days of actual surveillance as off-set term in the model. Longitudinal prevalence of disease will be calculated for each individual as the percentage of actual surveillance days with illness. All continuous variables (longitudinal prevalence, body iron status, mean and total weight and height gain) will be analysed using linear mixed models using cluster, household and child as random effects to account for clustered observations. Mixed effects logistic regression analysis will be used to evaluate binary outcomes (anemia, iron deficiency and iron-deficiency anemia), using cluster, household and child as random effects. All models will include the following fixed effects as co-variates: child's sex, socio-economic status, and baseline values. Non-normal distributed values will be log-transformed. P-values of < 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Living in one of the selected intervention and non-intervention villages
* Between 6 months and 11.99 months old at the day of recruitment
* Have not yet been provided with MNPs as part of the project interventions
* Free of chronic conditions that may impact their health
* Caregivers do not plan to migrate out of the study area
* Caregivers have provided written informed consent for this additional safety component

Exclusion Criteria:

* Children who are severely malnourished (Wt/Ht Z-score < -3 SD) will be referred to treatment and excluded from the safety component
* Children with a chronic disease and/or chronic use of medications
* Children who are severe anemic (Hb< 70 g/L)

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2356 (Actual)
Dates: Start 2015-03; Primary Completion 2016-05 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Anemia | Baseline and Endline
  Hemoglobin <110g/L
% of new acute diarrhea episodes (>3 loose stools/day) per 52 surveillance weeks | Up to one year
  Morbidity from diarrhea (prevalence and incidence rate)

SECONDARY OUTCOMES:
Iron status | Baseline and Endline
  Iron status measured by iron deficiency (ID) and iron deficiency anemia (IDA). ID defined as serum ferritin (SF) concentration <12µg/L. IDA defined as hemoglobin <110g/L with SF<12µg/L.
% of new respiratory infection episodes (cough and/or difficult breathing with or without fever, accompanied by rapid breathing and chest in drawing) per 52 surveillance weeks | Up to one year
  Morbidity from any types of flu (flu,common cold or cough)-prevalence and incidence rate
Prevalence of Fever | Up to one year
  Body temperature >37.5 degree Centigrade per 52 surveillance weeks
Growth | Up to one year
  Change in height-for-age Z-score (HAZ), weight-for-length Z-score (WHZ), and weight-for-age Z-score (WAZ)

CONTACTS AND LOCATIONS:
Overall Officials: Saskia JM Osendarp, PhD, Study Chair — Micronutrient Initiative; Inge D Brouwer, PhD, Study Director — Wageningen University
Locations (1):
- Ethiopian Public Health Institute, Addis Ababa, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hayes RJ, Bennett S. Simple sample size calculation for cluster-randomized trials. Int J Epidemiol. 1999 Apr;28(2):319-26. doi: 10.1093/ije/28.2.319. PMID 10342698
- [Background] Zimmermann MB, Chassard C, Rohner F, N'goran EK, Nindjin C, Dostal A, Utzinger J, Ghattas H, Lacroix C, Hurrell RF. The effects of iron fortification on the gut microbiota in African children: a randomized controlled trial in Cote d'Ivoire. Am J Clin Nutr. 2010 Dec;92(6):1406-15. doi: 10.3945/ajcn.110.004564. Epub 2010 Oct 20. PMID 20962160
- [Background] Erhardt JG, Estes JE, Pfeiffer CM, Biesalski HK, Craft NE. Combined measurement of ferritin, soluble transferrin receptor, retinol binding protein, and C-reactive protein by an inexpensive, sensitive, and simple sandwich enzyme-linked immunosorbent assay technique. J Nutr. 2004 Nov;134(11):3127-32. doi: 10.1093/jn/134.11.3127. PMID 15514286
- [Background] Cook JD, Flowers CH, Skikne BS. The quantitative assessment of body iron. Blood. 2003 May 1;101(9):3359-64. doi: 10.1182/blood-2002-10-3071. Epub 2003 Jan 9. PMID 12521995
- [Derived] Samuel A, Osendarp SJM, Feskens EJM, Lelisa A, Adish A, Kebede A, Brouwer ID. Gender differences in nutritional status and determinants among infants (6-11 m): a cross-sectional study in two regions in Ethiopia. BMC Public Health. 2022 Feb 26;22(1):401. doi: 10.1186/s12889-022-12772-2. PMID 35219315